CLINICAL TRIAL: NCT05228236
Title: Comparing the Effects of Plant Based Protein vs. Whey Protein on Performance and Body Composition of Futsal Players
Brief Title: Plant Based Protein and Whey Protein: Effects on Body Composition and Performance
Acronym: 4BettPro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bettery S.A. (Industry)
Responsible Party: Principal Investigator, Filipe Teixeira, Innovation Manager, Bettery S.A.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BetteryLifeLab4BP
Record Dates: First submitted 2022-01-13; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Protein Supplementation
Keywords: Plant-based Protein; Body composition; Physical Performance; Biochemical Health Markers; Supplementation
MeSH Terms: interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant based protein (Experimental)
  Interventions: Dietary Supplement: Plant based protein
- Whey Protein (Experimental)
  Interventions: Dietary Supplement: Whey protein

INTERVENTIONS:
Dietary Supplement: Plant based protein — A single dose of ~30 g of a plant-based protein blend was ingested 30-60 min after physical practice in training days or 30-60 min before bedtime in resting days.
  Arms: Plant based protein
Dietary Supplement: Whey protein — A single dose of ~30 g of whey protein was ingested 30-60 min after physical practice in training days or 30-60 min before bedtime in resting days.
  Arms: Whey Protein

SUMMARY:
This study aimed to investigate the effects of a newly developed plant-based protein blend regarding health and safety, body composition, and performance on healthy and physically active adult individuals, specifically team sports athletes. A randomized, double-blind, controlled trial was used to compare the effects of the plant-based protein versus whey protein, after an 8-week supplementation protocol, on body composition, biochemical markers, muscle strength and power, as well as aerobic performance in male futsal players. The working hypothesis is that this special blend of plant-based protein will be equivalent to whey protein, not only regarding body composition and performance, but also insofar as health and safety at the biochemical and physiological level.

DETAILED DESCRIPTION:
A randomized, double-blind, controlled trial was performed to investigate health and safety following supplementation with a newly developed plant-based protein blend and to compare the effects of this plant-based protein versus whey protein, after an 8-week supplementation protocol, on body composition and performance. Prior to intervention, volunteers' general health and ability to participate in the study were assessed. The study involved 50 male futsal players currently engaged in a training program and competing. Before engaging the 8-week supplementation protocol, participants underwent measurements of body composition, strength and power, and aerobic performance, as well as a full profile of biochemical health markers, and assessment of food and fluid intake. Evaluations were repeated after 4 weeks, for follow up and to detect potential compliance issues, and after 8 weeks of supplementation. Assessments took place in the morning (starting at 7:00 a.m.) after an overnight fast, except for the performance tests, which were performed following consumption of a standard, meal replacement bar.

Anthropometry and Body Composition - Wearing minimal clothing and no shoes, participants had their weight and height measured on a scale and stadiometer (Seca, Hamburg, Germany), respectively. Body composition, namely bone mineral content, fat mass and fat free mass, were evaluated by dual energy X-ray absorptiometry (DXA) (Horizon Wi, Hologic, Waltham, USA) and skeletal muscle through the evaluation of the muscle thickness of the rectus femoris by ultrasonography (model WED-180 HL, Shenzhen,China). Total body water and its intra and extracellular compartments were estimated from whole body resistance (R) and reactance (Xc), measured through bioelectrical impedance analysis (BIA), using a single frequency device of 50 kHz (BIA-101, RJL/Akern Systems, Firenze, Italy). From the raw R and Xc data, the phase angle was additionally determined, using the Akern Software.

Muscle Strength and Power, and Aerobic Performance - Strength was assessed using the handgrip strength test, as well as the back squat and bench press 1 repetition maximum (1 RM). The handgrip strength test was used to evaluate the maximal isometric force of the muscles of the hand and forearm. Using a portable hand dynamometer (JAMAR, Sammons Preston, Bolingbrook, IL, USA), participants were assessed for both hands alternately, in a stand-up position. The maximal force generated out of 3 attempts was considered for analysis. Additionally, muscle strength was evaluated by 1RM back squat and bench press in a Multipower machine, using a velocity-based training device (Vitruve Encoder, Madrid, Spain). Muscle power was assessed during maximal cycling (Wingate test) and jumping movements. During the Wingate test, participants were instructed to cycle (Monark 894 Peak Bike, Vansbro, Sweden) against a predetermined resistance (7.5% body weight), as fast as possible, for 30 seconds. Vertical jumps, namely the squat jump, countermovement jumps using both legs and single legs, as well as the Abalakov countermovement jump, were performed on a multicomponent force platform (Chronojump Boscosystem, Barcelona, Spain) interfaced with a computer. The best out of 3 attempts was also considered for analysis of this methodology. Aerobic performance was assessed by VO2peak and maximal aerobic speed (MAS), determined using a breath-by-breath gas analyzer (Quark, Cosmed, Italy) in an incremental test performed on a treadmill (Axelero, MEDEN-INMED, Koszalin, Poland). After 3 minutes of warm-up at 5 km/h, participants began the test at 6 km/h and 2% inclination. Each minute, the speed increased 1 km/h until volitional exhaustion. The VO2peak was considered the highest 30 sec average value of VO2 and MAS, the speed at the last completed stage.

All tasks were performed by the participants with direct supervision of sport scientists and/or exercise physiologists, with prior knowledge of the methodologies, and experience handling the equipments and corresponding softwares.

Biochemical Markers - For biochemical health markers, saliva and whole blood, in EDTA tubes, were collected per the standard protocols. . From whole blood, plasma was separated when necessary. Blood measurements included hematocrit, glucose, C-reactive protein (CRP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), creatine kinase (CK), and creatinine, using spectrophotometry techniques in an automated equipment (Vario Photometer II DP310, Diglobal Gmbh, Berlin, Germany). Saliva was collected for cortisol evaluation in Enzyme-Linked Immunosorbent Assay (ELISA) commercial kits (Salimetrics, PA, USA).

Nutritional Assessment - Following extensive verbal and written instructions, diet control and food patterns were characterized using 3-day food records (2 non-consecutive weekdays and 1 weekend day). Participants were instructed to maintain their dietary pattern for the 8 weeks of the study. Energy, macronutrient, and micronutrient intake were quantified using a dietary analysis software (Nutritics Research Edition (v5.09), Dublin, Ireland).

Randomization and Supplementation - Eligible participants were assigned to one of the two arms of the study using a covariate adaptive randomization procedure considering the covariates age, handgrip strength, whole body fat-free mass, and whole-body fat mass percentage. The investigator responsible for the sample randomization and supplements distribution was not directly involved in participants' eligibility interview or data collection. The supplementation protocol was similar for both the plant-based and whey protein, with the uptake of a single dose of ~30 g occurring 30-60 min after physical practice on training days or 30-60 min before bedtime on rest days. Supplementation compliance was assessed by questionnaire at the end of weeks 4 and 8.

Sample Size Justification - Previous, similar studies showed no differences between the abovementioned supplements regarding the analyzed variables of interest. In cases where there are no differences between the arms of the study, an effect size does not exist, so a power analysis is not a valid approach. As our hypothesis is that there will be no difference between the newly developed plant-based protein blend and whey protein, we can consider a non-inferiority trial and, therefore, our sample size can be similar to that of previous studies. Additionally, despite the time course of muscle hypertrophy not being exactly known, an 8-week intervention would be considered the minimum timeline for true hypertrophy to be detectable/measurable after 6-8 weeks of resistance training (using medical imageology i.e., ultrasound). Furthermore, it has been reported that to detect hypertrophy differences following supplementation with proteins of different quality, the number of subjects needed should be in the range of at least 25 per group. We have chosen to go with a robust approach. Therefore, our proposed sample size is of 25 participants per group.

Statistics - All statistical analyses are being carried out using IBM SPSS Statistics (Version 25.0, NY, IBM). Basic descriptive data were run to characterize the study participants. All variables were checked for normality, using Kolmogorov-Smirnov test. Participants were assigned to either a plant-based protein (n = 25) or animal protein group (n = 25), based on handgrip strength, age, fat mass or fat-free mass using a stratified random assignment. Independent Sample T tests will be applied to compare means between supplementation groups, at baseline. Time and time-by-group interactions will be evaluated by repeated-measures ANOVA. The equality of the matrix of variance and sphericity will be explored with the Levene F test and Mauchly's test, respectively. Overall significance level for α will be set at p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Subjects currently engaged in a Futsal training program in a competition team, currently engaged in practice for at least 1 year and at least 3 times per week.

Exclusion Criteria:

* Individuals taking any type of drug (including anabolic steroids), medicines or supplements that may enhance body composition or performance, 3 months prior to the beginning of the trial.
* Clinical diagnose of a disease that might compromise tolerance to the supplements or influence body composition or performance.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Body composition parameter - change in fat free mass (FFM) | Baseline, week 4 and week 8
  FFM (kg) was assessed by dual energy X-ray absorptiometry
Body composition parameter - change in fat mass (FM) | Baseline, week 4 and week 8
  FM (%) was assessed by dual energy X-ray absorptiometry
Body composition parameter - change in muscle thickness | Baseline, week 4 and week 8
  muscle thickness of the rectus femoris (mm) was assessed by ultrasonography
Body composition parameter - change in body water | Baseline, week 4 and week 8
  total body water, intracellular water and extracellular water (L) were assessed by bioelectrical impedance analysis
Performance parameter - change in strength | Baseline, week 4 and week 8
  Maximal isometric forearm strength (N) was assessed using a handgrip dynamometer
Performance parameter - change in maximum strength | Baseline, week 4 and week 8
  Maximum strength (kg) was predicted from 1-RM in back squat and bench press exercises using a Multipower machine withVitruve technology
Performance parameter - change in peak power | Baseline, week 4 and week 8
  Muscle power (Watt) was assessed with a supramaximal cycling test on cycle ergometer
Performance parameter - change in jump height | Baseline, week 4 and week 8
  Vertical jump height (cm) was assessed on a multicomponent force platform interfaced with the Chronojump software
Aerobic performance - change in Oxygen uptake | Baseline, week 4 and week 8
  VO2peak (mL.kg-1.min-1) was assessed using breath-by-breath gas analyzer in an incremental test performed on a treadmill
Aerobic performance - change in Oxygen uptake | Baseline, week 4 and week 8
  Maximal aerobic speed (km/h) was assessed in an incremental test performed on a treadmill
biochemical health markers - change in cortisol | Baseline, week 4 and week 8
  Salivary cortisol was assessed using spectrophotometry techniques in an automated equipment.
biochemical health markers - change in creatinine | Baseline, week 4 and week 8
  plasma creatinine was assessed using spectrophotometry techniques in an automated equipment.
biochemical health markers - change creatine kinase | Baseline, week 4 and week 8
  plasma creatine kinase was assessed using spectrophotometry techniques in an automated equipment.
biochemical health markers - change in glucose | Baseline, week 4 and week 8
  plasma glucose was assessed using spectrophotometry techniques in an automated equipment.
biochemical health markers - change in C reactive protein | Baseline, week 4 and week 8
  plasma C Reactive Protein was assessed using spectrophotometry techniques in an automated equipment.
biochemical health markers - change in Aspartate Aminotransferase | Baseline, week 4 and week 8
  plasma Aspartate Aminotransferase was assessed using spectrophotometry techniques in an automated equipment.
biochemical health markers - change in alanine aminotransferase | Baseline, week 4 and week 8
  Plasma alanine aminotransferase was assessed using spectrophotometry techniques in an automated equipment.

SECONDARY OUTCOMES:
Body composition parameter - change in phase angle | Baseline, week 4 and week 8
  Phase angle (degree) was assessed by bioelectrical impedance analysis
Body composition parameter - change of visceral fat | Baseline, week 4 and week 8
  Visceral fat (kg) was assessed by dual energy X-ray absorptiometry

CONTACTS AND LOCATIONS:
Locations (1):
- Bettery S.A., Oeiras, Porto Salvo, Portugal

IPD SHARING:
Plan to Share IPD: No